CLINICAL TRIAL: NCT00018291
Title: Specific Interventions for Agitation in Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AGCG-005-00S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Dementia; Agitated Behavior; Behavioral disturbance
MeSH Terms: conditions — Alzheimer Disease; Dementia; Psychomotor Agitation; Mental Disorders | interventions — Risperidone; Gabapentin

INTERVENTIONS:
Drug: Risperidone
Drug: Gabapentin

SUMMARY:
This study is aimed at investigating specific pharmacological interventions in the treatment of the disruptive, agitated behavior associated with Alzheimer's patients. In addition, it is hoped that specific clinical profiles will be found to predict which treatment is most effective for these particular patients.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is the most common cause of dementia, the fourth leading cause of death, and has enormous economic and emotional costs for caregivers of patients. Most of the patients with AD develop disruptive, agitated behaviors at some point during the ailment that are a common catalyst for placement in long-term care settings where they represent more than half of all the residents. Disruptive behaviors create stress for both staff and patients in long-term care settings, reduce patient quality of life because of excess use of physical restraints, and drain the financial resources of the facilities. This study proposes to design specific interventions designed to decrease disruptive, agitated behavior in patients with AD residing in long-term care facilities. This 12-week study will assess the efficacy of two pharmacological agents, an atypical neuroleptic (risperidone) and an anticonvulsant and mood stabilizer (gabapentin) while identifying moderators of differential treatment response to the two drugs. Specifically, this study aims to randomize 130 patients with AD who are manifesting agitated disruptive behavior, into two groups of 65 patients each, with one group receiving risperidone and the other gabapentin. There are two main hypotheses: 1) Patients in both of the treatment groups will manifest different overall group decreases in ratings of disruptive, agitated behavior; and 2) Measurable, clinical characteristics will identify subgroups of subjects with differential treatment response to the two medications. The two variables to be considered as moderators are as follows: a) Patients with higher psychosis ratings will manifest greater responsivity to risperidone compared to gabapentin, and b) Patients with high levels of affective lability will manifest greater responsivity to gabapentin compared to risperidone.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of probable AD according to DSM-IV, which show high agreement with NINCDS-ADRDA criteria (McKhann et al., 1984); kappa = 0.81 (Chui et al., in press).
2. At least a two-week history of two or more agitated behaviors from the Agitation Screening Inventory (a shortened version of the 24-item Revised Memory and Behavior Problem Checklist) (RMBPC; Teri at al., 1992), occurring at least once weekly, and rated by the caregiver or nursing staff as at least moderately distressing.
3. Not planning a change in living situation or placement during the investigational period.
4. Stability (of dose and type) of medications for nonexcluded concurrent medical conditions (i.e. thyroid disease, anemia, cardiac disease) for four weeks prior to baseline.
5. Ability to ingest oral medications and participate in all scheduled evaluations.
6. A sixth grade education or a work history sufficient to exclude mental retardation.
7. 50 years of age or older.
8. Medically acceptable for experimental drugs as confirmed by physical evaluation and laboratory tests.
9. Modified Hachinski Scale score of 4 or less.

Exclusion Criteria

1. Neurological diagnoses other than AD which affect cognitive function. These include Parkinson?s Disease, tumors, hydrocephalus, history of significant trauma, and seizure disorder).
2. A diagnosis of delirium by the Confusion Assessment Method (CAM, Inouye et al., 1990).
3. A diagnosis of dementia related to infection with human immunodeficiency virus (HIV) or amnestic disorder, as defined by DSM-IV.
4. Known hypersensitivity to risperidone or gabapentin.
5. Alcohol or drug abuse within the past year.
6. Serious, unstable medical illnesses (e.g., unstable angina, poorly controlled diabetes mellitus, labile hypertension)
7. Any medical problem that would cause or exacerbate agitated behaviors (including unstable thyroid dysfunction, electrolyte disturbances, urinary tract infection, fecal impaction, respiratory disease complicated by hypoxia or hypercapnia, etc.)
8. Any psychotropic medications or other medications which may cause or exacerbate agitated behavior. Patients taking these medications may participate in the study if the drugs can be successfully discontinued during the washout period and the remainder of the study, and if after discontinuation they still meet inclusion criteria for the investigation. Excluded medications include: antipsychotics; antidepressants; anxiolytics; CNS stimulants; anti convulsants; and sedative hypnotics.
9. Significantly abnormal laboratory findings.
10. Significantly abnormal EKG findings.
11. Conditions such as blindness, deafness, or other disability that may prevent the patient from participating in the study.
12. Current participation in any other investigational drug study or treatment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto VA Health Care System, Menlo Park, California, United States